CLINICAL TRIAL: NCT03683979
Title: An Investigation of the Short-term Impact of Interpretation Bias Modification Training on Anger Symptoms, Reactive Aggression, and Attentional Biases Toward Anger-related Stimuli
Brief Title: The Impact of Interpretation Bias Modification Training on Anger and Reactive Aggression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Monique Tremblay, Monique D Tremblay, M.A Ryerson University, Toronto Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Anger Study 1
Record Dates: First submitted 2018-09-22; First posted 2018-09-25 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Anger
Keywords: Reactive aggression; High trait anger; Cognitive bias modification; Interpretation bias modification

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interpretation bias modification program (Experimental): Participants in this arm will complete a computer-based training program two times in the lab. Participants will complete the first training session in the lab during their initial visit and they will return to the lab one week later to complete the second session.
  Interventions: Behavioral: Interpretation Bias Modification
- Control training program (Sham Comparator): Participants in this arm will complete a sham training program two times in the lab. The program will look similar in length and design to the experimental training program, but the content of the program will remain affectively neutral. As in the experimental condition, participants will complete the first training session in the lab during their initial visit and they will return to the lab one week later to complete the second session.
  Interventions: Behavioral: Control Training Program

INTERVENTIONS:
Behavioral: Interpretation Bias Modification — A computer based interpretation bias modification program that aims to reinforce neutral interpretations of ambiguous social situations.
  Arms: Interpretation bias modification program
Behavioral: Control Training Program — A sham training program that is similar in design and delivery to the experimental training condition.
  Arms: Control training program

SUMMARY:
Difficulties with anger control are reported in a number of psychological conditions and are associated with social problems, such as dating violence and workplace violence. High trait anger is a personality construct characterized by elevations in the frequency, duration, and intensity of anger episodes. However, the cognitive processes contributing to high trait anger are still poorly understood. This study will examine the effectiveness of a computer-based cognitive bias modification (CBM) program designed to target hostile interpretations associated with high trait anger.

DETAILED DESCRIPTION:
High trait anger is a personality construct characterized by elevations in the frequency, duration, and intensity of anger episodes. According to the Integrative Cognitive Model (ICM) of anger, three cognitive processes jointly contribute to an individual's level of trait anger and reactive aggression: hostile attributions, ruminative attention, and effortful control processes. Specifically, individuals high in trait anger are more prone to interpret ambiguous situations as hostile; are more likely to ruminate about anger-related events; and have a more limited capacity to employ control processes when they become angry.

One means of evaluating unconscious biases that has become increasingly popular is cognitive bias modification (CBM). CBM programs are computerized training paradigms, which aim to train more adaptive cognitive biases by repeatedly exposing participants to an experimental contingency between an emotional stimulus and a response.Previous researchers have begun to investigate the impact of CBMs targeting cognitive control and hostile attribution bias in relation to anger. However, these studies have been conducted exclusively in samples reporting low trait anger.

This study will examine the effectiveness of a short-term interpretation bias modification program (CBM-I) on hostile attribution biases and reactive aggression in a sample of undergraduate students eporting high trait anger.

ELIGIBILITY:
Inclusion Criteria:

1. Students scoring 22 or higher on the Trait Anger Scale.

Exclusion Criteria:

1. Reports currently receiving psychological treatment or counseling for anger.
2. Reports changes in psychiatric medication within the last month.
3. Endorsement of current psychosis or bipolar disorder symptoms.
4. Indicates poor English language proficiency.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
State-Trait Anger Expression Inventory 2nd Edition | Administered two times over the course of one week. Changes will be examined from visit 1 (before CBM training program) to visit 2 (after CBM training program).
  A self-report measure of the experience of anger.
Interpretation Bias Assessment | Administered two times over the course of one week. Changes will be examined from visit 1 (before CBM training program) to visit 2 (after CBM training program).
  A computer-based measure of hostile interpretation bias involving ambiguous social scenarios.

SECONDARY OUTCOMES:
Anger Rumination Scale | Administered two times over the course of one week. Changes will be examined from visit 1 (before CBM training program) to visit 2 (after CBM training program).
  A self-report measure of the degree to individuals focus on experiences with anger. The scale is comprised of four subscales, angry after thoughts (e.g., "Whenever I experience anger, I keep thinking about it for a while"), angry memories (e.g., "I re-enact the anger episode in my mind after it has happened"), understanding causes (e.g., "When someone provokes me, I keep wondering why this should have happened to me"), and thoughts of revenge (e.g. "I have difficulty forgiving people who have hurt me."). Participants will be asked to read each item and rate it in terms of how well it reflects their experience on a 4-point scale from 1 ("almost never") to 4 ("almost always"). Totals for each sub scale will be summed to produce a total score (range: 19-76), with higher scores indicating a greater propensity for rumination.
Social Information Processing-Attribution and Emotional Response Questionnaire | Administered two times over the course of one week. Changes will be examined from visit 1 (before CBM training program) to visit 2 (after CBM training program).
  A self-report measure of evaluate social information processing biases associated with hostile attribution bias.
Word Sentence Association Paradigm-Hostility | Administered two times over the course of one week. Changes will be examined from visit 1 (before CBM training program) to visit 2 (after CBM training program).
  A behavioural measure of hostile attribution biases involving hostile and non-hostile words.
Depression and Anxiety Stress Scale-21 | Administered two times over the course of one week. Changes will be examined from visit 1 (before CBM training program) to visit 2 (after CBM training program).
  A self-report measure of depression, anxiety, and stress symptoms. A self-report measure of depression, anxiety, and stress symptoms.Items are summed for each subscale to create subscale totals (i.e., depression, anxiety, and stress), with higher scores reflecting more severe emotional distress. Symptom score ranges include: normal (0-4), mild (5-6), moderate (7-10), severe (11-13), and extremely severe (14+).
Dot Probe | Administered two times over the course of one week. Changes will be examined from visit 1 (before CBM training program) to visit 2 (after CBM training program).
  A behavioural measure of attentional bias towards angry faces.
Reactive-Proactive Aggression Questionnaire | Administered two times over the course of one week. Changes will be examined from visit 1 (before CBM training program) to visit 2 (after CBM training program).
  A self-report measure of an individual's propensity for reactive aggression.
Taylor Aggression Paradigm | Administered one time over the course of one week. Participants will be exposed to the paradigm following the second training session.
  A behavioural measure of reactive aggression.

CONTACTS AND LOCATIONS:
Locations (1):
- Ryerson University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The results of this study will be disseminated through conference presentations and journal publications. Anonymized aggregate participant data may be made available upon request to a publishing journal or individual research group. However, research groups interested in accessing anonymized data will be required to submit a proposal detailing their intended use of the data. Their qualifications will be reviewed based on their proposal and CVs. Individual research groups approved for access will be required to agree to not attempt to re-identify participants, not further distribute data, and not use the data for purposes other than specified in their original proposal. No individual data will be shared.

REFERENCES:
- [Background] Hawkins KA, Cougle JR. Effects of interpretation training on hostile attribution bias and reactivity to interpersonal insult. Behav Ther. 2013 Sep;44(3):479-88. doi: 10.1016/j.beth.2013.04.005. Epub 2013 Apr 19. PMID 23768674
- [Background] Wilkowski BM, Robinson MD. The cognitive basis of trait anger and reactive aggression: an integrative analysis. Pers Soc Psychol Rev. 2008 Feb;12(1):3-21. doi: 10.1177/1088868307309874. Epub 2007 Dec 18. PMID 18453470